CLINICAL TRIAL: NCT00644306
Title: Comparison of Melphalan-Prednisone (MP) to MP Plus Thalidomide in the Treatment of Newly Diagnosed Very Elderly Patients (> 75 Years) With Multiple Myeloma
Acronym: IFM 01/01
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: survival advantage demonstrated
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Hulin Cyrille, Intergroupe Francophone du Myélome (IFM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University Hospital, Nancy
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Newly Diagnosed, Multiple Myeloma
Keywords: Multiple Myeloma, very elderly patients, thalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; AP protocol 2; Melphalan; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): 12 cycles every 6 weeks :melphalan 0.2 mg/kg day 1 to 4, prednisone 2 mg/kg/d day 1 to 4 plus placebo 100mg/d continuously for 18 months
  Interventions: Drug: Thalidomide; Drug: melphalan, prednisone
- B (Active Comparator): 12 cycles every 6 weeks :melphalan 0.2 mg/kg day 1 to 4, prednisone 2 mg/kg/d day 1 to 4 plus thalidomide 100mg/d continuously for 18 months
  Interventions: Drug: melphalan, prednisone, thalidomide

INTERVENTIONS:
Drug: Thalidomide — 100 mg/day continuously for 18 months
  Arms: A
Drug: melphalan, prednisone — 12 cycles every 6 weeks :melphalan 0.2 mg/kg day 1 to 4, prednisone 2 mg/kg/d day 1 to 4 plus placebo 100mg/d continuously for 18 months
  Other Names: Alkeran, cortancyl
  Arms: A
Drug: melphalan, prednisone, thalidomide — 12 cycles every 6 weeks :melphalan 0.2 mg/kg day 1 to 4, prednisone 2 mg/kg/d day 1 to 4 plus thalidomide 100mg/d continuously for 18 months
  Other Names: Alkeran, cortancyl
  Arms: B

SUMMARY:
In multiple myeloma, combination chemotherapy with melphalan plus prednisone has been usedsince the 1960s and is regarded as the standard of care in very elderly patients. We assess whether the addition of thalidomide at 100 mg/day to this combination would improve survival.

ELIGIBILITY:
Inclusion Criteria:

* Stage II or III multiple myeloma according to Durie and Salmon criteria, patients older than 75 years, previously untreated patients.

Exclusion Criteria:

* Prior history of another neoplasm (except basocellular cutaneous or cervical epithelioma)
* Primary or associated amyloïdosis
* World Health organisation performance index of at least 3
* Significant renal insufficiency with creatinine serum levels of 5.0 mg per deciliter or more
* Cardiac or hepatic dysfunction
* Cerebral circulatory insufficiency
* Absolute contraindication to corticosteroids
* Peripheral neuropathy clinically significant
* History of venous thrombosis during the last 6 months
* HIV or hepatitis B or C positivity
* Patients who had geography, social, or psychological conditions which might prevent adequate follow-up.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 232 (Actual)
Dates: Start 2002-04; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
overall Survival | May 2007

SECONDARY OUTCOMES:
Progression Free Survival | May 2007
Response rates | May 2007
Safety | May 2007

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille Hulin, MD, Principal Investigator — Hematology CHU Nancy and Intergroupe Francophone du Myelome (IFM)
Locations (1):
- CHU Nancy - Brabois, rue du morvan, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Background] Facon T, Mary JY, Hulin C, Benboubker L, Attal M, Pegourie B, Renaud M, Harousseau JL, Guillerm G, Chaleteix C, Dib M, Voillat L, Maisonneuve H, Troncy J, Dorvaux V, Monconduit M, Martin C, Casassus P, Jaubert J, Jardel H, Doyen C, Kolb B, Anglaret B, Grosbois B, Yakoub-Agha I, Mathiot C, Avet-Loiseau H; Intergroupe Francophone du Myelome. Melphalan and prednisone plus thalidomide versus melphalan and prednisone alone or reduced-intensity autologous stem cell transplantation in elderly patients with multiple myeloma (IFM 99-06): a randomised trial. Lancet. 2007 Oct 6;370(9594):1209-18. doi: 10.1016/S0140-6736(07)61537-2. PMID 17920916